CLINICAL TRIAL: NCT00239434
Title: Comparison of 18 mg of Tiotropium Inhalation Capsules Once Daily and Atrovent Metered Dose Inhaler (2 Puffs of 20 mg, Four Times Daily) in a Double-Blind, Double-dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Comparison of 18g of Tiotropium Inhalation Capsules Once Daily and Atrovent Metered Dose Inhaler (2 Puffs of 20g, 4 Times Daily) in a Double-Blind, Double-Dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.245
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: tiotropium inhalation powder capsule
Drug: ipratropium bromide Metered Dose Inhaler

SUMMARY:
The objective of this study is to compare the bronchodilator efficacy and safety of once daily dosing of tiotropium inhalation capsules (18 ?g) and Atrovent? MDI (2 puffs of ipratropium bromide 20 ?g four times daily) in patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, parallel group study to compare the bronchodilator efficacy and safety of tiotropium inhalation capsules and Atrovent? MDI in patients with chronic obstructive pulmonary disease (COPD).

Following an initial screening visit, patients will enter a 2-week baseline period. Patients who successfully complete this phase will be randomized into the double-blind portion of the study in which they will receive tiotropium once daily (morning) or Atrovent? four times daily for 4 weeks. Pulmonary function testing will be conducted just prior (i.e. 5 minutes before) to the start of therapy at Visit 2 (i.e. randomization visit after completion of the 2-week run-in period) and at 30, 60, 120 and 180 minutes post-dosing. Pulmonary function testing will be repeated at the same time intervals after 14 days of therapy (visit 3) and at the end of therapy.

Those patients taking theophylline, will be questioned about their last theophylline intake in order to ensure adherence to the washout requirements.

Vital signs will be measured in conjunction with the pulmonary function tests. Adverse events will be recorded throughout the entire run-in and treatment period.

Study Hypothesis:

The null hypothesis is that there is no difference in mean response between tiotropium and Atrovent. The alternative hypothesis is that there is a difference in mean response between tiotropium and Atrovent.

Comparison(s):

The primary pulmonary function variable will be FEV1 (Forced Expiratory Volume in one second) and trough FEV1 response at the end of the four week treatment period, i.e. visit 4, will be the primary efficacy endpoint.

Trough FEV1 is defined as FEV1 at the end of the dosing interval (for tiotropium at approximately 24 hours post treatment administration). On test days (Visits 3 and 4) it is measured by the PFT just prior to dosing. Trough FEV1 response is defined as change from baseline in trough FEV1. Baseline FEV1 is defined as FEV1 measured just prior to first dosing in the morning of randomization visit (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a diagnosis of chronic obstructive pulmonary disease according to the following criteria:

   Patients must have relatively stable airway obstruction with an FEV1 ? 65% of predicted normal and FEV1 70% of FVC.

   Predicted normal values will be based on the following formula. Males: FEV1 pred.(L) = height2(m) x (-0.016 x age(year) + 1.823) Females: FEV1 pred.(L) = height2(m) x (-0.012 x age(year) + 1.4427)
2. Male or female patients 40 years of age or older.
3. Patients must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year.
4. Patients must be able to perform pulmonary function tests as required in the protocol.
5. Patients must be able to inhale medication from the HandiHaler device and should have a good technique of inhaling aerosol administered from an MDI.
6. All patients must sign an Informed Consent Form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications.

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded.
3. All patients with a SGOT and SGPT twice the normal range, bilirubin 150% or creatinine 125% of the normal range will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these subjects.
4. Patients with a recent history (i.e. one year or less) of myocardial infarction.
5. Patients with a recent history (i.e. three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
6. Patients with regular use of daytime oxygen therapy.
7. Patients with known active tuberculosis.
8. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed.
9. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
10. Patients who have undergone pulmonary resection.
11. Patients with an upper respiratory tract infection in the past 6 weeks prior to the Screening Visit (=Visit 1) or during the baseline period of 2-weeks (run-in period).
12. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other component of the inhalation capsule delivery system or the MDI.
13. Patients with known symptomatic prostatic hyperplasia or bladder neck obstruction.
14. Patients with known narrow-angle glaucoma.
15. Patients who are being treated with cromolyn sodium or nedocromil sodium.
16. Patients who are being treated with antihistamines.
17. Patients using oral corticosteroid medication at unstable (i.e. less than 6 weeks on a stable dose) or at a dose in excess of the equivalent 10 mg of prednisone per day or 20 mg every other day.
18. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices, or diaphragm).
19. Patients with a history of asthma, allergic rhinitis or atopy or who have a blood total eosinophil count >= 400 per µl (males) or >= 320 per µl (females). A repeat eosinophil count will not be conducted in these patients.
20. Patients with a history and/or active alcohol or drug abuse.
21. Patients who have taken an investigational drug one month or six half-lives (whichever is greater) prior to the Screening Visit (=Visit 1).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-06; Study Completion 2004-03

PRIMARY OUTCOMES:
Trough FEV1 response: change from baseline trough FEV1 (visit 2) at visit 4

SECONDARY OUTCOMES:
Trough FEV1 response at visit 3 Average FEV1 (AUC0-3) response (change from baseline) for the 3 hours post drug administration Trough FVC response Average FVC (AUC0-3) response (as defined for FEV1) 5. Amount of rescue medication 6. Patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (6):
- China (6):
  - People Hospital of Beijing University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - 1st Hospital of Guangzhou Medical College, Guangzhou
  - Zhongshan Hospital of Fudan University, Shanghai
  - Shanghai 1st People Hospital, Shanghai
  - 1st Hospital of Chinese Medical University, Shenyang